CLINICAL TRIAL: NCT04634357
Title: An Open-Label, Dose Escalation, Phase I/II Clinical Trial of ET140203 T Cells in Pediatric Subjects With Relapsed/Refractory Hepatoblastoma (HB), Hepatocellular Neoplasm-Not Otherwise Specified (HCN-NOS), or Hepatocellular Carcinoma (HCC)
Brief Title: ET140203 T Cells in Pediatric Subjects With Hepatoblastoma, HCN-NOS, or Hepatocellular Carcinoma
Acronym: ARYA-2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eureka Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETUS20AFPAR123
Record Dates: First submitted 2020-11-04; First posted 2020-11-18 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hepatoblastoma; Hepatocellular Carcinoma (HCC); Liver Neoplasms; Metastatic Liver Cancer; Liver Cancer; HEMNOS
Keywords: Relapsed/Refractory Hepatoblastoma (HB); Pediatric; Hepatocellular Neoplasm-Not Otherwise Specified (HCN-NOS); Hepatocellular Carcinoma (HCC); Liver Cancer; T-cell therapy; Metastatic Liver Cancer; Liver neoplasms; HEMNOS
MeSH Terms: conditions — Hepatoblastoma; Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ET140203 T Cells (Experimental): ET140203 Autologous T Cells
  Interventions: Drug: ET140203 T Cells

INTERVENTIONS:
Drug: ET140203 T Cells — Biological/Vaccine: ET140203 autologous T-cell product
  Autologous T cells transduced with lentivirus encoding an ET140203 expression construct

SUMMARY:
Open-label, dose escalation, multi-center, Phase I/II clinical trial to assess the safety/tolerability and determine the recommended Phase II Dose (RP2D) of ET140203 T-cells in pediatric subjects who are AFP-positive/HLA-A2-positive and have relapsed/refractory HB, HCN-NOS, or HCC.

DETAILED DESCRIPTION:
The trial starts with a dose escalation phase. A traditional dose escalation model (3+3) design will be used to determine the recommended phase II dose (RP2D). Subjects will then be treated at the RP2D in the expansion phase of the trial.

Following treatment, tumor response assessments will be performed at Months 1, 3, 6, 9, 12, 18, and 24. At each tumor response assessment visit, imaging will be performed (triphasic CT Scan) and used for response evaluation. Serum AFP levels will also be measured at each tumor response assessment visit.

The active assessment phase of the study will continue for 2 years. Subjects will be followed for 15 years post-treatment for assessment of treatment safety and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed HB, HCN-NOS, or HCC with serum AFP >100ng/mL at the time of screening and following the most recent line of therapy.
2. Disease reoccurrence after remission following initial standard-of care (SOC) treatment (i.e., relapse) or failure of response to SOC treatment (i.e., refractory).
3. Age ≥ 1 year and ≤ 21 years.
4. Molecular Human Leukocyte Antigen (HLA) class I allele typing that confirms subject carries at least one HLA-A2 allele.
5. Life expectancy of > 4 months per the Investigator's opinion.
6. Lansky or Karnofsky Performance Scale ≥ 70.
7. For enrollment to the dose-finding cohort, subjects must have at least one (1) lesion ≥ 5 mm in diameter or two (2) or more lesions ≥ 3 mm in diameter. For the dose-expansion cohort, subjects must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
8. Child-Pugh score of A6 or better.
9. Adequate organ function.

Exclusion Criteria:

1. Recurrent HB who are candidates for complete surgical resection (e.g., isolated pulmonary relapse amendable to pulmonary metastasectomy).
2. Pre-existing illness including heart failure, uncontrolled pulmonary disease not cancer-related, or psychiatric illness/social situation that would limit compliance with study requirements.
3. Active, uncontrolled systemic bacterial, fungal, or viral infection. Subjects with Human Immunodeficiency Virus (HIV), hepatitis B, or hepatitis C are eligible provided their infection is being treated and the viral load is controlled.
4. Any known active malignancy (other than HB, HCN-NOS, or HCC).
5. Pregnant or lactating women.
6. Received the following within two (2) weeks of leukapheresis or within two (2) weeks of conditioning chemotherapy: cytotoxic chemotherapy, radiation, other anti-cancer therapies (including immunotherapeutic agents), immunosuppressive therapy, or systemic corticosteroids at doses greater than 5 mg/day of prednisone or equivalent doses of other corticosteroids. (Note: Topical and inhaled corticosteroids in standard doses and physiological replacement doses of corticosteroids for adrenal insufficiency are allowed).
7. Concurrently receiving other investigational agents, biological, chemical, or radiation therapies, while participating in the study.
8. Contraindication for receipt of conditioning chemotherapeutic agents including Fludarabine and Cyclophosphamide.
9. Active autoimmune disease requiring systemic immunosuppressive therapy.
10. Compromised circulation in the main portal vein, hepatic vein, or vena cava due to partial or complete obstruction which, in the opinion of the Investigator, would make the subject unsuitable for the study.
11. History of organ transplant.
12. HB, HCN-NOS, or HCC involving greater than 50% of the liver (volumetric).

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rates of adverse events (AEs) after infusion of ET140203 T cells | 28 days
  Safety of ET140203 T cells as assessed by the number of adverse events (AEs) after infusion
Severity rates of adverse events (AEs) after infusion of ET140203 T cells | 28 days
  Safety of ET140203 T cells as assessed by the severity of adverse events (AEs) after infusion.
Incidence rates of dose limiting toxicities (DLTs) after infusion of ET140203 T cells | 28 days
  Tolerability of ET140203 T cells after infusions assessed by committee review of dose limiting toxicities (DLTs)
The recommended phase 2 dose (RP2D) regimen of ET140203 T cell therapy primarily based on DLT | Up to 2 years
  The RP2D will be determined by the study Dose Escalation Committee (DEC) and primarily based on DLTs.

SECONDARY OUTCOMES:
Assess the efficacy of ET140203 T cells in pediatric subjects with relapsed/refractory HB, HCN-NOS, or HCC | Up to 2 years
  Response rate will be assessed by radiographic scans and assessed according to RECIST criteria.
Determine the pharmacokinetics of ET140203 T cells after infusion. | Up to 2 years
  Assess the expansion and persistence of ET140203 T cells circulating in blood over time.

CONTACTS AND LOCATIONS:
Overall Officials: Pei Wang, PhD, Study Director — Eureka Therapeutics Inc.
Locations (2):
- United States (2):
  - UCSF Benioff Children's Hospitals, San Francisco, California
  - Dana-Farber/Boston Children's Cancer and Blood Disorders Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No